CLINICAL TRIAL: NCT04741698
Title: Propranolol for Prolonged Labor: A Randomized Controlled Trial (PRO-Labor Trial)
Brief Title: Propranolol for Protracted Labor
Acronym: PRO-Labor
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DDD# 604829
Record Dates: First submitted 2021-01-15; First posted 2021-02-05 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Labour;Obstructed; Labor Dystocia
MeSH Terms: conditions — Dystocia | interventions — Propranolol; propranolol CR

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propranolol 2mg IV (Active Comparator): At the time of labor dystocia, patients randomized to the treatment arm of propranolol will receive a one-time administration of IV 2mg propranolol in pre-mixed syringes prepared by the pharmacy.
  The propranolol IV administration recommended in clinical practice guidelines is 1 mg IV over 1 minute. Therefore, total administration time will be 2 minutes.
  Interventions: Drug: Propranolol
- No intervention (No Intervention): At the time of labor dystocia, patients randomized to the placebo arm will not receive any intervention

INTERVENTIONS:
Drug: Propranolol — Propranolol 2mg IV
  Other Names: Propranolol Hydrochloride; Inderal; Inderal LA; InnoPran XL; Hemangeol
  Arms: Propranolol 2mg IV

SUMMARY:
Induction of labor is one of the most common procedures performed on labor and delivery. In the United States, more than 20 percent of pregnant women undergo an induction of labor [1].

There is data from small, randomized studies that demonstrates the effectiveness of propranolol, a non-selective beta-blocker, for labor augmentation. This literature suggests a decrease in the amount of time to delivery and a possible reduction in cesarean section rates when propranolol is used in conjunction with oxytocin for induction of labor compared to oxytocin alone [2-8].

Alpha- and beta-adrenergic receptors have been identified in the human myometrium. Propranolol has been shown in studies to enhance uterine contractions and may be a useful tool in this population of women. Therefore, the purpose of this study is to assess whether the administration of propranolol at time of labor dystocia reduces time to delivery.

DETAILED DESCRIPTION:
All cervical ripening will be performed in the labor and delivery unit; continuous fetal heart rate and uterine activity will be monitored in all patients. Cervical dilation is assigned by admitting physicians. Sonography will be performed to document fetal presentation.

At the time of prolonged labor, patients meeting inclusion criteria and no exclusion criteria will be consented. There will be no monetary incentives for participation.

Patients will be randomized to either Propranolol 2mg of IV or expectant management at the time of induction. Maternal vitals will be collected per standard labor management.

Episodes of uterine activity that are deemed excessive by the physician will be treated with a standard combination of maneuvers that included a change in maternal position, oxygen administration, and terbutaline 250 µg subcutaneously. Persistent abnormal fetal heart rate patterns resulted in intervention by removing the patient from the study. Urgent cesarean delivery is defined as a cesarean delivery performed during the ripening process for abnormal fetal heart rate that did not respond to standard maneuvers.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* full term (≥37 weeks) gestations determined by routine obstetrical guidelines
* singleton gestation in cephalic presentation
* Intact membranes
* Bishop score of ≤6 and cervical dilation ≤2cm

Exclusion Criteria:

* Preterm gestation
* Diabetes requiring insulin in labor: given the potential risk of neonatal hypoglycemia in the neonate
* multiparous women
* Any cardiac condition for which β blockade is contraindicated (cardiogenic shock, sinus bradycardia, and greater than first degree heart block)
* Known hypersensitivity to propranolol
* Maternal bradycardia (HR <60bpm)
* Severe preeclampsia: as patients will be receiving magnesium and possibly labetalol for hypertension control
* Systolic blood pressure <90 mmHg, or diastolic blood pressure <50 mmHg
* Receiving other beta blocker
* Moderate or severe asthma: as this is a contraindication to beta blocker use
* Any contraindication to a vaginal delivery
* fetal demise
* Multifetal gestation
* major fetal anomaly
* prior uterine surgery, previous cesarean section
* women with HIV, hepatitis C, hepatitis B, and women with medical conditions requiring an assisted second stage
* Additional exclusion criteria were as follows: category 3 fetal heart rate tracing, hemolysis elevated liver enzymes and low platelets (HELLP) syndrome or eclampsia, growth restriction <10th percentile (based on Hadlock growth curves) with reversal of flow in umbilical artery Doppler studies, and growth restriction <5th percentile with elevated, absent, or reversal of flow in umbilical artery Doppler studies.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2022-06-11 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
time to delivery | Number of hours from induction to delivery of neonate; up to 72 hours.
  The primary outcome is time to delivery (hours) defined as time from initiation of induction method to delivery time, regardless of mode of delivery.

SECONDARY OUTCOMES:
cesarean delivery rate | At time of delivery
  rate of cesarean delivery
maternal length of stay | From time of admission to time of hospital discharge; an average of two days
  from time of admission to discharge
Maternal Bradycardia event | at time of delivery
  bradycardia alert during labor
Chorioamnionitis | At time of delivery
  defined by the presence of maternal fever ≥100·4°f in the presence of maternal or fetal tachycardia or fundal tenderness
neonatal admission to ICU | At time of delivery
  NICU admission
Severe respiratory distress syndrome | at time of delivery
  defined as intubation and mechanical ventilation for a minimum of 12 hours
neonatal sepsis | at time of delivery
  Culture proven-presumed neonatal sepsis
Neonatal blood transfusion | From time of delivery to time of hospital discharge; up to 6 weeks
  Neonatal blood transfusion
Hypoxic ischemic encephalopathy | through study completion, an average of 1 year
  neonatal HIE

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Gomez, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moghadam AD, Jaafarpour M, Khani A. Comparison effect of oral propranolol and oxytocin versus oxytocin only on induction of labour in nulliparous women (a double blind randomized trial). J Clin Diagn Res. 2013 Nov;7(11):2567-9. doi: 10.7860/JCDR/2013/5704.3613. Epub 2013 Nov 10. PMID 24392402
- [Background] Kashanian M, Fekrat M, Zarrin Z, Ansari NS. A comparison between the effect of oxytocin only and oxytocin plus propranolol on the labor (a double blind randomized trial). J Obstet Gynaecol Res. 2008 Jun;34(3):354-8. doi: 10.1111/j.1447-0756.2008.00790.x. PMID 18588611
- [Background] Pergialiotis V, Frountzas M, Prodromidou A, Prapa S, Perrea DN, Vlachos GD. Propranolol and oxytocin versus oxytocin alone for induction and augmentation of labor: a meta-analysis of randomized trials. Arch Gynecol Obstet. 2016 Apr;293(4):721-9. doi: 10.1007/s00404-015-3991-8. Epub 2015 Dec 22. PMID 26695642
- [Background] Pruyn SC, Phelan JP, Buchanan GC. Long-term propranolol therapy in pregnancy: maternal and fetal outcome. Am J Obstet Gynecol. 1979 Oct 15;135(4):485-9. doi: 10.1016/0002-9378(79)90436-8. PMID 573555
- [Background] Sanchez-Ramos L, Quillen MJ, Kaunitz AM. Randomized trial of oxytocin alone and with propranolol in the management of dysfunctional labor. Obstet Gynecol. 1996 Oct;88(4 Pt 1):517-20. doi: 10.1016/0029-7844(96)00223-2. PMID 8841209
- [Background] Meidahl Petersen K, Jimenez-Solem E, Andersen JT, Petersen M, Brodbaek K, Kober L, Torp-Pedersen C, Poulsen HE. beta-Blocker treatment during pregnancy and adverse pregnancy outcomes: a nationwide population-based cohort study. BMJ Open. 2012 Jul 19;2(4):e001185. doi: 10.1136/bmjopen-2012-001185. Print 2012. PMID 22815467
- [Background] Palomaki O, Uotila J, Tammela O, Kaila T, Lavapuro M, Huhtala H, Tuimala R. A double blind, randomized trial on augmentation of labour with a combination of intravenous propranolol and oxytocin versus oxytocin only. Eur J Obstet Gynecol Reprod Biol. 2006 Mar 1;125(1):44-9. doi: 10.1016/j.ejogrb.2005.06.016. Epub 2005 Jul 26. PMID 16051416